CLINICAL TRIAL: NCT02752035
Title: A Phase 3 Multicenter, Open-label, Randomized Study of ASP2215 (Gilteritinib), Combination of ASP2215 Plus Azacitidine and Azacitidine Alone in the Treatment of Newly Diagnosed Acute Myeloid Leukemia With FLT3 Mutation in Patients Not Eligible for Intensive Induction Chemotherapy
Brief Title: A Study of ASP2215 (Gilteritinib) by Itself, ASP2215 Combined With Azacitidine or Azacitidine by Itself to Treat Adult Patients Who Have Recently Been Diagnosed With Acute Myeloid Leukemia With a FLT3 Gene Mutation and Who Cannot Receive Standard Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-0201; 2015-001790-41 (EudraCT Number)
Expanded Access: NCT03070093 (Approved for marketing)
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia With FMS-like Tyrosine Kinase (FLT3) Mutation
Keywords: AML; ASP2215; Newly Diagnosed AML; gilteritinib; Acute Myeloid Leukemia (AML); FLT3
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Cohort: Gilteritinib + Azacitidine (AZA) (Experimental): Participants received 80 mg (2 tablets of 40 mg) of gilteritinib orally once daily for continuous 28-day cycles and 75 mg/m^2 of AZA daily via subcutaneous injection or intravenous infusion for 7 days of each 28-day treatment cycle. Depending on the safety cohort data ,the decision to initiate the randomized trial at the targeted dose was made. After the end of treatment period, participants were followed up for 30- day follow up period. Participants were allowed to enter the long-term follow-up period of up to 3 years for collection of subsequent AML treatment, EQ-5D-5L, remission status and survival (cause of death and date of death). Participants in long-term follow-up who were no longer receiving treatment were followed every 3 months for survival until the implementation of the final protocol version 13.0, at which time they were discontinued from the study, as further survival data were no longer needed.
  Interventions: Drug: gilteritinib; Drug: azacitidine
- Randomized Cohort: Gilteritinib + AZA (Experimental): Participants received 120 mg(3 tablets of 40 mg)of gilteritinib orally once daily for continuous 28-day cycles in combination with 75mg/m^2 of AZA daily via subcutaneous injection or IV infusion for 7days of each 28-day treatment cycle until the participant no longer received clinical benefit from therapy in the opinion of the investigator,unacceptable toxicity occurred,or the participant met another treatment discontinuation criterion.After the end of treatment period,participants were followed up for 30-day follow up period.Participants were allowed to enter the long-term follow-up period of up to 3 years for collection of subsequent AML treatment,EQ-5D-5L,remission status and survival (cause and date of death).Participants in long-term follow-up who were no longer receiving treatment were followed every 3months for survival until the implementation of the final protocol version 13.0, at which time they were discontinued from the study,as further survival data were no longer needed.
  Interventions: Drug: gilteritinib
- Randomized Cohort: AZA (Experimental): Participants received 75 mg/m^2 of AZA daily via subcutaneous injection or intravenous infusion for 7 days of each 28-day treatment cycle until the participant no longer received clinical benefit from therapy in the opinion of the investigator, unacceptable toxicity occurred or the participant met another treatment discontinuation criterion. After the end of treatment period, participants were followed up for 30- day follow up period. Participants were allowed to enter the long-term follow-up period of up to 3 years for collection of subsequent AML treatment, EQ-5D-5L, remission status and survival (cause of death and date of death). Participants in long-term follow-up who were no longer receiving treatment were followed every 3 months for survival until the implementation of the final protocol version 13.0, at which time they were discontinued from the study, as further survival data were no longer needed.
  Interventions: Drug: gilteritinib; Drug: azacitidine
- Randomized Cohort: Gilteritinib (Active Comparator): Participants received 120 mg (3 tablets of 40 mg) of gilteritinib orally once daily for continuous 28-day cycles until the participant no longer received clinical benefit from therapy in the opinion of the investigator, unacceptable toxicity occurred or the participant met another treatment discontinuation criterion. However, randomization to this arm was removed in protocol version 7.0. Participants previously randomized to this arm continued following treatment and assessments as outlined in the protocol.
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: gilteritinib — Tablet, oral
  Other Names: ASP2215
  Arms: Randomized Cohort: AZA; Randomized Cohort: Gilteritinib + AZA; Safety Cohort: Gilteritinib + Azacitidine (AZA)
Drug: azacitidine — Subcutaneous injection or intravenous infusion
  Arms: Randomized Cohort: AZA; Randomized Cohort: Gilteritinib; Safety Cohort: Gilteritinib + Azacitidine (AZA)

SUMMARY:
This was a clinical study for adult participants who were recently diagnosed with acute myeloid leukemia or AML. AML is a type of cancer. It is when bone marrow makes white blood cells that are not normal. These are called leukemia cells. Some participants with AML have a mutation, or change, in the FLT3 gene. This gene helps leukemia cells make a protein called FLT3. This protein causes the leukemia cells to grow faster.

For participants with AML who could not receive standard chemotherapy, azacitidine (also known as Vidaza®) was a current standard of care treatment option in the United States. This clinical study tested an experimental medicine called ASP2215, also known as gilteritinib. Gilteritinib worked by stopping the leukemia cells from making the FLT3 protein. This helped stop the leukemia cells from growing faster.

This study compared two different treatments. Participants were assigned to one of these two groups by chance: a medicine called azacitidine, also known as Vidaza®, or an experimental medicine gilteritinib in combination with azacitidine. There was a twice as much chance to receive both medicines combined than azacitidine alone. The clinical study may help show which treatment helps patients live longer.

DETAILED DESCRIPTION:
Participants considered an adult according to local regulation at the time of obtaining informed consent participated in the study.

Safety Cohort Prior to initiation of the randomized trial, 15 participants were enrolled to evaluate the safety and tolerability of ASP2215 given with azacitidine therapy in the study population.

Randomized Trial Approximately 250 participants were randomized in a 2:1 ratio to receive ASP2215 plus azacitidine (Arm AC) or azacitidine only (Arm C). Participants entered the screening period up to 14 days prior to the start of treatment. Participants administered treatment over 28-day cycles.

Earlier protocol versions included a 1:1:1 randomization ratio to receive Arm A: ASP2215, Arm AC: ASP2215 + azacitidine or Arm C: azacitidine. Participants previously randomized to Arm A continued following treatment and assessments as outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of obtaining informed consent.
* Subject has a diagnosis of previously-untreated AML according to World Health Organization (WHO) classification [Swerdlow et al, 2008] as determined by pathology review at the treating institution.
* Subject is positive for FLT3 mutation (internal tandem duplication [ITD] or tyrosine kinase domain [TKD] [D835/I836] mutation) (or for Korea only: ITD alone or ITD with concurrent TKD activating mutation) in bone marrow or whole blood as determined by central laboratory. Note: Only requirement of FLT3 mutation assessment by central laboratory is only applicable to the randomization portion of the study.
* Subject is ineligible for intensive induction chemotherapy by meeting at least 1 of the following criteria:

  * Subject is ≥ 65 years of age and ineligible for intensive induction chemotherapy.
  * Subject is ≥ 18 to 64 years of age and has any of the following comorbidities: [Ex-US Only]: Congestive heart failure (New York Heart Association {NYHA} class ≤ 3) or ejection fraction (Ef) ≤ 50%; [US Only]: Severe cardiac disorder e.g. congestive heart failure (New York Heart Association [NYHA] class ≤ 3) requiring treatment, ejection fraction ≤ 50%, or chronic stable angina; [Ex-US Only]: Creatinine > 2 mg/dL (177 µmol/L), dialysis or prior renal transplant; [US Only]: Creatinine clearance < 45 mL/min; ECOG performance status ≥ 2;
  * [Ex-US Only]: Known pulmonary disease with decreased diffusion capacity of lung for carbon monoxide (DLCO) and/or requiring oxygen ≤ 2 liters per minute; [US Only] Severe pulmonary disorder (e.g., diffusion capacity of lung for carbon monoxide [DLCO] ≤ 65% or forced expiratory volume in the first second [FEV1] ≤ 65%); Prior or current malignancy that does not require concurrent treatment; Subject has received a cumulative anthracycline dose above 400 mg/m2 of doxorubicin (or cumulative maximum dose of another anthracycline). Any other comorbidity incompatible with intensive chemotherapy must be reviewed and approved by the Medical Monitor during screening and before randomization.
* Subject must meet the following criteria as indicated on the clinical laboratory tests:

  * Serum AST and ALT ≤ 3.0 x Institutional upper limit of normal (ULN)
  * Serum total bilirubin ≤ 1.5 x Institutional ULN
  * Serum potassium ≥ Institutional lower limit of normal (LLN)
  * Serum magnesium ≥ Institutional LLN Repletion of potassium and magnesium levels during the screening period is allowed.
* Subject is suitable for oral administration of study drug.
* Female subject is eligible to participate if female subject is not pregnant and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP); OR
  * WOCBP agrees to follow the contraceptive guidance starting at screening and continue throughout the study period, and for at least 180 days after the final study drug administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 60 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 180 days after the final study drug administration.
* Male subject with female partners of childbearing potential must agree to use contraception as detailed in Contraception Requirements, starting at screening and continue throughout the study period, and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject was diagnosed as acute promyelocytic leukemia (APL).
* Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has received previous therapy for AML, with the exception of the following:

  * Emergency leukapheresis
  * Hydroxyurea
  * Preemptive treatment with retinoic acid prior to exclusion of APL ≤ 7 days
  * Growth factor or cytokine support
  * Steroids
* Subject has clinically active central nervous system leukemia.
* Subject has been diagnosed with another malignancy that requires concurrent treatment (with the exception of hormone therapy limited to those therapies that prevent recurrence and/or spread of cancer) or hepatic malignancy regardless of need for treatment.
* Subject requires treatment with concomitant drugs that are strong inducers of cytochrome P450 CYP3A/P-glycoprotein (P-gp).
* Subject requires treatment with concomitant drugs that are strong inhibitors or inducers of P-gp with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject requires treatment with concomitant drugs that target serotonin 5-hydroxytryptamine receptor 2B (5HT2BR) or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the subject.
* Subject has congestive heart failure classified as New York Heart Association Class IV.
* Subject with mean Fridericia-corrected QT interval (QTcF) > 480 ms at screening based on central reading.
* Subject with a history of Long QT Syndrome at screening.
* [Ex-US Only]: Subject has known pulmonary function tests with diffusion capacity of lung for carbon monoxide (DLCO) ≤ 50%, forced expiratory volume in the first second (FEV1) ≤ 60%, dyspnea at rest or requiring oxygen or any pleural neoplasm (Transient use of supplemental oxygen is allowed.)
* Subject has active hepatitis B or C or other active hepatic disorder.

  * Subjects with positive hepatitis B surface antigen (HBsAg) or detectable hepatitis B DNA are not eligible.
  * Subjects with negative HBsAg, positive hepatitis B core antibody and negative hepatitis B surface antibody will be eligible if hepatitis B DNA is undetectable.
  * Subjects with antibodies to hepatitis C virus will be eligible if hepatitis C RNA is undetectable
* Subject has any condition which makes the subject unsuitable for study participation, including any contraindications of azacitidine.
* Subject has a known or suspected hypersensitivity to ASP2215, azacitidine or any components of the formulations used.
* [US Only]: Subject is ≥ 65 to 74 years of age, suitable for and willing to receive intensive induction chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (111):
- United States (12):
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Louis University Cancer Center - Hematology/Oncology, St Louis, Missouri
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - GHS Cancer Institute, Greenville, South Carolina
  - LDS Hospital, Salt Lake City, Utah
- Australia (3):
  - Site AU61004, Liverpool, New South Wales
  - Site AU61008, Adelaide, South Australia
  - Site AU61007, Geelong, Victoria
- Belgium (3):
  - Site BE32007, Brussels, Brussels Capital
  - Site BE32003, Brussels, Bruxelles-Capitale, Region de
  - Site BE32006, Ghent
- Canada (4):
  - Site CA15009, Edmonton, Alberta
  - Site CA15011, Toronto, Ontario
  - Site CA15002, Toronto, Ontario
  - Site CA15006, Montreal, Quebec
- France (14):
  - Site FR33003, Nîmes, Gard
  - Site FR33002, Pessac, Gironde
  - Site FR33015, Rouen, Haute-Normandie
  - Site FR33019, Montpellier, Herault
  - Site FR33018, Rennes, Ille-et-Vilaine
  - Site FR33001, Nantes, Loire-Atlantique
  - Site FR33023, Valenciennes, Nord
  - Site FR33013, Pierre-Bénite, Rhone
  - Site FR33017, Le Mans, Sarthe
  - Site FR33012, Poitiers, Vienne
  - Site FR33009, Angers
  - Site FR33020, Bayonne
  - Site FR33004, Lille
  - Site FR33006, Lille
- Germany (9):
  - Site DE49002, Tübingen, Baden-Wurttemberg
  - Site DE49007, München, Bavaria
  - Site DE49005, Frankfurt am Main, Hesse
  - Site DE49012, Braunschweig, Lower Saxony
  - Site DE49004, Hanover, Lower Saxony
  - Site DE49015, Rostock, Mecklenburg-Vorpommern
  - Site DE49009, Halle, Saxony-Anhalt
  - Site DE49003, Berlin
  - Site DE49011, Stuttgart
- Italy (10):
  - Site IT39009, Ancona
  - Site IT39015, Bologna
  - Site IT39012, Florence
  - Site IT39004, Milan
  - Site IT39007, Monza
  - Site IT39001, Napoli
  - Site IT39014, Novara
  - Site IT39006, Palermo
  - Site IT39005, Pavia
  - Site IT39011, San Giovanni Rotondo
- Japan (26):
  - Site JP81018, Anjo, Aichi-ken
  - Site JP81007, Nagoya, Aichi-ken
  - Site JP81027, Matsuyama, Ehime
  - Site JP81021, Fukuyama, Hiroshima
  - Site JP81031, Sapporo, Hokkaido
  - Site JP81033, Sapporo, Hokkaido
  - Site JP81015, Kobe, Hyōgo
  - Site JP81034, Hitachi, Ibaraki
  - Site JP81023, Kanazawa, Ishikawa-ken
  - Site JP81001, Isehara, Kanagawa
  - Site JP81032, Yokohama, Kanagawa
  - Site JP81012, Sendai, Miyagi
  - Site JP81011, Kurashiki, Okayama-ken
  - Site JP81029, Shibuya-ku, Tokyo
  - Site JP81014, Shinagawa-ku, Tokyo
  - Site JP81035, Chiba
  - Site JP81008, Fukuoka
  - Site JP81024, Gifu
  - Site JP81005, Kumamoto
  - Site JP81016, Kyoto
  - Site JP81004, Nagasaki
  - Site JP81017, Nagasaki
  - Site JP81030, Osaka
  - Site JP81036, Osaka
  - Site JP81026, Tokushima
  - Site JP81019, Toyama
- Poland (4):
  - Site PL48003, Lublin, Lublin Voivodeship
  - Site PL48004, Warsaw, Masovian Voivodeship
  - Site PL48002, Opole, Opole Voivodeship
  - Site PL48001, Olsztyn, Warmian-Masurian Voivodeship
- South Korea (9):
  - Site KR82003, Namdong, Incheon Gwang'yeogsiv
  - Site KR82013, Seoul, Seoul Teugbyeolsi
  - Site KR82006, Seoul, Seoul Teugbyeolsi
  - Site KR82002, Seoul, Seoul Teugbyeolsi
  - Site KR82001, Ulsan, Ulsan Gwang'yeogsi
  - Site KR82014, Busan
  - Site KR82010, Hwasun-gun
  - Site KR82015, Seongnam-si
  - Site KR82012, Seoul
- Spain (9):
  - Site ES34007, Palma de Mallorca, Balearic Islands
  - Site ES34003, Oviedo, Principality of Asturias
  - Site ES34008, Barcelona
  - Site ES34004, Barcelona
  - Site ES34010, Barcelona
  - Site ES34009, Barcelona
  - Site ES34002, Cáceres
  - Site ES34013, Madrid
  - Site ES34005, Valencia
- Taiwan (7):
  - Site TW88604, Kaohsiung City
  - Site TW88605, Kwei Shan Hsiang
  - Site TW88602, Tainan
  - Site TW88609, Tainan
  - Site TW88601, Taipei
  - Site TW88608, Taipei
  - Site TW88610, Taipei
- Site GB44007, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Wang ES, Montesinos P, Minden MD, Lee JH, Heuser M, Naoe T, Chou WC, Laribi K, Esteve J, Altman JK, Havelange V, Watson AM, Gambacorti-Passerini C, Patkowska E, Liu S, Wu R, Philipose N, Hill JE, Gill SC, Rich ES, Tiu RV. Phase 3 trial of gilteritinib plus azacitidine vs azacitidine for newly diagnosed FLT3mut+ AML ineligible for intensive chemotherapy. Blood. 2022 Oct 27;140(17):1845-1857. doi: 10.1182/blood.2021014586. PMID 35917453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed, FMS-like tyrosine kinase 3 (FLT3)-mutated acute myeloid leukemia (AML) not eligible for intensive induction were enrolled.
Pre-assignment Details: Prior to randomized cohort, participants were enrolled for safety cohort to evaluate safety and tolerability of gilteritinib given with azacitidine therapy.
Groups:
- Randomized Cohort: Gilteritinib + AZA: Participants received 120 mg (3 tablets of 40 mg) of gilteritinib orally once daily for continuous 28-day cycles in combination with 75 mg/m^2 of AZA daily via subcutaneous injection or intravenous infusion for 7 days of each 28-day treatment cycle until the participant no longer received clinical benefit from therapy in the opinion of the investigator, unacceptable toxicity occurred or the participant met another treatment discontinuation criterion.After the end of treatment period, participants were followed up for 30- day follow up period. Participants were allowed to enter the long-term follow-up period of up to 3 years for collection of subsequent AML treatment, EQ-5D-5L, remission status and survival (cause of death and date of death). Participants in long-term follow-up who were no longer receiving treatment were followed every 3 months for survival until the implementation of the final protocol version 13.0, at which time they were discontinued from the study, as further survival data were no longer needed.
Period: Safety Cohort: Approximately 5 Years
Arm/Group | Safety Cohort: Gilteritinib + Azacitidine (AZA) | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Started | 15 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 0 | 0 | 0
Not completed — Miscellaneous | 2 | 0 | 0 | 0
Not completed — Disease relapse | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Death | 5 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Randomization: Approximately 3 Years
Arm/Group | Safety Cohort: Gilteritinib + Azacitidine (AZA) | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Started | 0 | 89 | 57 | 22
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 89 | 57 | 22
Not completed — Miscellaneous | 0 | 7 | 4 | 1
Not completed — Disease Relapse | 0 | 22 | 16 | 6
Not completed — Physician Decision | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 14 | 7 | 4
Not completed — Lack of Efficacy | 0 | 4 | 14 | 0
Not completed — Death | 0 | 25 | 13 | 4
Not completed — Adverse Event | 0 | 14 | 2 | 6
Period: Long-term Follow-up: up to 3 Years
Arm/Group | Safety Cohort: Gilteritinib + Azacitidine (AZA) | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Started | 5 | 33 | 34 | 10
Completed | 0 | 0 | 0 | 0
Not Completed | 5 | 33 | 34 | 10
Not completed — Withdrawal by Subject | 0 | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Death | 5 | 26 | 30 | 10
Not completed — Miscellaneous | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as the intention to treat set, which consisted of participants who were randomized and were used for efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Cohort: Gilteritinib + Azacitidine (AZA) | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib | Total
Number analyzed (Participants) | 15 | 89 | 57 | 22 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.3 (5.6) | 77.1 (5.7) | 76.9 (5.2) | 78.5 (4.2) | 77.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 40 | 27 | 10 | 85
  Male | 7 | 49 | 30 | 12 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 14 | 75 | 46 | 18 | 153
  Unknown or Not Reported | 1 | 12 | 7 | 3 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data reported for Race.
  Participants
    Race: White | 11 | 53 | 33 | 9 | 106
    Race: Asian | 3 | 25 | 15 | 10 | 53
    Race: Unknown | 1 | 11 | 8 | 2 | 22
    Race: Other | 0 | 0 | 1 | 1 | 2
Age group per Interactive Response Technology (IRT) [Count of Participants; unit: Participants] — IRT is a system used in clinical trials to manage randomization, treatment allocation, and trial supply logistics.
  Participants
    < 75 years | 6 | 27 | 15 | 4 | 52
    >= 75 years | 9 | 62 | 42 | 18 | 131
FMS-like tyrosine kinase 3 (FLT3) mutation type [Count of Participants; unit: Participants] — FLT3 is a receptor tyrosine kinase that is expressed almost exclusively in the hematopoietic compartment.
  Participants
    Internal Tandem Duplication (ITD) Alone | 10 | 70 | 46 | 17 | 143
    Tyrosine Kinase Domain (TKD) (D835/I836) Alone | 3 | 16 | 9 | 2 | 30
    ITD with TKD (D835/I836) | 1 | 3 | 2 | 3 | 9
    Others (unknown/missing/negative) | 1 | 0 | 0 | 0 | 1
Cytogenetic risk status [Count of Participants; unit: Participants] — The cytogenetic risk status was categorized as Favorable [Core binding factor: inv(16) or t(16;16) or t(8;21). Other cytogenetic abnormalities in addition to these do not alter better risk status], Intermediate [Normal cytogenetics, +8 alone, t(9;11), Other non-defined cytogenetic abnormality], or Unfavorable [Complex (≥ 3 clonal chromosomal abnormalities), Monosomal karyotype, -5, 5q-, -7, 7q-, 11q23 - non t(9;11), inv(3), t(3;3), t(6;9)]
  Participants
    Favorable | 0 | 2 | 0 | 0 | 2
    Intermediate | 11 | 63 | 40 | 17 | 131
    Unfavorable | 1 | 9 | 6 | 0 | 16
    Others (unknown, missing) | 3 | 15 | 11 | 5 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause. For a participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact. Kaplan-Meier (KM) estimates was used for analysis.
Time Frame: From the date of randomization until the date of death from any cause ( maximum duration up to 79 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
months | 9.82 [8.11 to 13.17] | 9.23 [4.34 to 12.55] | 5.24 [2.46 to 15.18]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Stratification factors were age group per IRT, risk groups and baseline FLT3 mutation status, with potential of strata pooling; Test type: Superiority; p = 0.523, Log Rank; Hazard Ratio (HR) = 0.870, 95% CI 2-sided [0.570 to 1.329] — Based on Cox proportional hazards model

2. Secondary Outcome: Event-free Survival (EFS)
Description: EFS: time from the date of randomization until the date of documented relapse from Complete Remission (CR), treatment failure(failing to achieve CR within 6 cycles of treatment) or death from any cause, whichever occurred first. CR: bone marrow(BM) regenerating normal hematopoietic cells, morphologically leukemia-free state, absolute neutrophil count (ANC) ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being red blood cell (RBC) and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. Relapse: reappearance of leukemic blasts >2% in the peripheral blood/≥ 5% myeloblasts in the BM unattributable to any other cause/new/reappearance of extramedullary leukemia.
Time Frame: From the date of randomization until the date of documented relapse from CR, treatment failure or death from any cause, whichever occurred first (up to 39.7 months)
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
months | 0.03 [NA to NA] — Lower and upper limits of the 95% confidence interval were not estimable due to insufficient number of participants with events. | 0.03 [NA to NA] — Lower and upper limits of the 95% confidence interval were not estimable due to insufficient number of participants with events. | 0.03 [0.03 to 2.46]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.787, Log Rank; Hazard Ratio (HR) = 0.940, 95% CI 2-sided [0.635 to 1.393] — Based on Cox proportional hazards model

3. Secondary Outcome: Percentage of Participants With Best Response
Description: Best response for a participant was defined as the best measured response (in the order of CR, CR with Incomplete Platelet Recovery (CRp), CR with Incomplete Hematologic Recovery (CRi), and treatment failure) from all post-baseline visits. CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. CRp: achieved CR except incomplete platelet recovery (< 100 × 10^9/L). CRi: achieved CR except incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence not required.
Time Frame: From the date of randomization until the date of death from any cause (up to 57 months)
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
percentage of participants
  CR | 25.8 | 17.5 | 9.1
  CRp | 6.7 | 0 | 18.2
  CRi | 29.2 | 10.5 | 27.3

4. Secondary Outcome: Completed Remission (CR) Rate
Description: CR rate: number of participants who achieved the best response of CR divided by the number of participants in the analysis population. Participants with unknown or missing response, or who provided no information on response at the end of treatment were included in the denominator when calculating rates. CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent(1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods.
Time Frame: From the date of randomization until the date of death from any cause (approximately 49.7 months)
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
percentage of participants | 25.8 | 17.5 | 9.1
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.249, Cochran-Mantel-Haenszel — Based on stratified Cochran-Mantel-Haenszel test. Stratification factor was age group per interactive response technology; Treatment Difference = 8.2, 95% CI 2-sided [-6.5 to 23.0]

5. Secondary Outcome: CRc Rate
Description: CRc rate was defined as participants with best response of (CR + CRp + CRi) divided by the number of participants in the analysis population. Participants were classified as: CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. CRp: achieved CR except incomplete platelet recovery (< 100 × 10^9/L). CRi: achieved CR except incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence not required. Percentage of participants with CRc was reported.
Time Frame: From the date of randomization until the date of death from any cause (approximately 54.5 months)
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
percentage of participants | 61.8 | 28.1 | 54.5
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 33.3, 95% CI 2-sided [16.6 to 50.0]

6. Secondary Outcome: Complete Remission With Partial Hematologic Recovery (CRh)
Description: CRh was defined as the response at a post baseline visit as CRh having bone marrow myeloblast count < 5%, partial hematologic recovery ANC ≥ 0.5 x 10^9/L and platelets ≥ 50 x 10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood must be ≤ 2% or missing. CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. Percentage of participants with CRh was reported.
Time Frame: From the date of randomization until the date of death from any cause (up to 49.7 months)
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
percentage of participants | 10.1 | 1.8 | 22.7
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 8.5, 95% CI 2-sided [-0.1 to 17.1]

7. Secondary Outcome: CR/CRh Rate
Description: CR/CRh rate: number of participants who achieved CR or CRh divided by the number of participants in the analysis population. CR/CRh: CR/CRh if it fulfilled criteria for CR or CRh at the visit. CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. CRh: response at a post baseline visit as CRh having bone marrow myeloblast count < 5%, partial hematologic recovery ANC ≥ 0.5 x 10^9/L and platelets ≥ 50 x 10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood must be ≤ 2% or missing. Percentage of participants with CR/CRh was reported.
Time Frame: From the date of randomization until the date of death from any cause (up to 49.7 months)
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 89 | 57 | 22
percentage of participants | 36.0 | 19.3 | 31.8
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.032, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 16.7, 95% CI 2-sided [1.1 to 32.4]

8. Secondary Outcome: Percentage of Participants With Transfusion Conversion Rate
Description: Transfusion conversion rate was defined as the number of participants who were transfusion dependent at baseline period but became transfusion independent at post-baseline period divided by the total number of participants who were transfusion dependent at baseline period.
Time Frame: From baseline up to 57 months
Population: FAS population included participants who were transfusion dependent at baseline period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 73 | 38 | 18
percentage of participants | 35.6 [24.7 to 47.7] | 44.7 [28.6 to 61.7] | 61.1 [35.7 to 82.7]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.340, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = -9, 95% CI 2-sided [-29.8 to 11.0]

9. Secondary Outcome: Percentage of Participants With Transfusion Maintenance Rate
Description: Transfusion maintenance rate was defined as the number of participants who were transfusion independent at baseline period and remained transfusion independent post-baseline period divided by the total number of participants who were transfusion independent at baseline period.
Time Frame: From baseline up to 57 months
Population: FAS population included participants who were transfusion independent at baseline period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 3 | 2 | 2
percentage of participants | 100.0 [29.2 to 100.0] | 50.0 [1.3 to 98.7] | 50.0 [1.3 to 98.7]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.221, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Treatment Difference = 50, 95% CI 2-sided [-61.0 to 100.0]

10. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS: time from the date of first CRc (CR + CRp + CRi) until the date of documented relapse (excluding relapse from PR) or death for participants who achieved CRc. CR: BM regenerating normal hematopoietic cells, morphologically leukemia-free state, ANC ≥1 × 10^9/L, platelet count ≥100 × 10^9/L, normal marrow differential with <5% myeloblast counts, missing/≤2% peripheral blood blast counts and being RBC and platelet transfusion independent (1 week without RBC and platelet transfusion prior to the disease assessment). No evidence of extramedullary leukemia and Auer rods. CRp: achieved CR except incomplete platelet recovery (< 100 × 10^9/L). CRi: achieved CR except incomplete hematological recovery with residual neutropenia < 1 x 10^9/L with or without complete platelet recovery. RBC and platelet transfusion independence not required. CRc: fulfilled criteria for CR, CRp or CRi. Based on KM estimates.
Time Frame: From first day of achieving first CRc to the first day of confirmed relapse/death (up to 54.5 months)
Population: FAS population included participants who had achieved CRc.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 55 | 16 | 12
months | 7.16 [6.01 to 12.52] | 8.08 [2.46 to 14.09] | 3.20 [0.89 to 6.87]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.592, Log Rank; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.451 to 1.580] — Based on Cox proportional hazards model adjusting age group per IRT

11. Secondary Outcome: Duration of Remission
Description: Duration of remission included CRc, CR, CRh, CR/CRh, and response duration [CRc + PR]. Duration of CRc, CR, CRh: the time from the date of first CRc until the date of first documented relapse for participants who achieved CRc, CR, and CRh, respectively. CR/CRh: fulfilled criteria for CR or CRh at the visit. CRh: marrow blasts <5%, ANC ≥0.5×10^9/L, platelets ≥50×10^9/L, not meeting CR criteria. PR: If marrow myeloblasts between <5% and 25% and ≤2% or missing peripheral blood blast and a decrease from baseline of at least 50% in the marrow myeloblasts and no evidence of extramedullary leukemia, the response was classified as PR. If marrow myeloblasts <5% and ≤2% or missing peripheral blood blast and no evidence of extramedullary leukemia, the response was classified as PR even with Auer rods.
Time Frame: From first day of achieving first response to the first day of confirmed relapse/death (up to 56.4 months)
Population: FAS population with available data was analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 61 | 21 | 16
months
  Duration of CR/CRh: number analyzed (Participants) | 32 | 11 | 7
  Duration of CR/CRh | 19.94 [6.93 to NA] — Median and upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival. | 8.08 [0.95 to 8.57] | 2.83 [1.87 to 5.95]
  Duration of CR: number analyzed (Participants) | 23 | 10 | 2
  Duration of CR | 25.10 [7.39 to NA] — Upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival. | 8.25 [0.95 to NA] — Upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival. | NA [NA to NA] — Median, lower and upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival.
  Duration of CRc: number analyzed (Participants) | 55 | 16 | 12
  Duration of CRc | 12.52 [6.77 to NA] — Upper limit of confidence interval was not estimable due to an insufficient number of events to determine 50% survival. | 8.25 [2.10 to 14.09] | 3.65 [0.89 to 7.39]
  Duration of CRh: number analyzed (Participants) | 9 | 1 | 5
  Duration of CRh | 6.77 [1.35 to 6.93] | 8.08 [NA to NA] — Lower and upper limit of 95% confidence interval was not estimable due to insufficient number of participants. | 2.83 [1.87 to 5.95]
  Duration of response | 7.92 [3.98 to 18.40] | 7.62 [0.95 to 9.23] | 3.65 [0.95 to 6.87]
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Analysis reported for duration of CR/CRh; Test type: Superiority; p = 0.300, Log Rank; Hazard Ratio (HR) = 0.573, 95% CI 2-sided [0.198 to 1.658] — Based on Cox proportional hazards model adjusting age group per IRT
Statistical Analysis 2: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Analysis reported for duration of CR; Test type: Superiority; p = 0.171, Log Rank; Hazard Ratio (HR) = 0.411, 95% CI 2-sided [0.113 to 1.504] — Based on Cox proportional hazards model adjusting age group per IRT
Statistical Analysis 3: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Analysis reported for duration of CRc; Test type: Superiority; p = 0.383, Log Rank; Hazard Ratio (HR) = 0.691, 95% CI 2-sided [0.295 to 1.620] — Based on Cox proportional hazards model adjusting age group per IRT
Statistical Analysis 4: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Analysis reported for duration of CRh; Test type: Superiority; p = 0.998, Log Rank; Hazard Ratio (HR) = 999, 95% CI 2-sided [lower limit 0.001] (Upper limit of 95% confidence interval was not estimable due to insufficient number of participants.) — Based on Cox proportional hazards model adjusting age group per IRT
Statistical Analysis 5: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Analysis reported for duration of response; Test type: Superiority; p = 0.174, Log Rank; Hazard Ratio (HR) = 0.628, 95% CI 2-sided [0.321 to 1.229] — Based on Cox proportional hazards model adjusting age group per IRT

12. Secondary Outcome: Change From Baseline in Brief Fatigue Inventory (BFI)
Description: The BFI was a tool to assess fatigue severity and impact on daily function in cancer participants over 24 hours. It included 9 items. A global fatigue score was computed by averaging the scores of the 9 items measured on the numeric rating scale. Scores were calculated if ≥5 of 9 items were answered. A higher score indicates a higher degree of fatigue. The first 3 rate fatigue from 0 (no fatigue) to 10 (worst imaginable), with higher scores indicating worse outcomes. The remaining 6 assess how fatigue interferes with daily activities from 0 (no interference) to 10 (completely interferes). A global fatigue score (0-10) was the average of all items, with higher scores indicating worse fatigue. Overall BFI score is reported.
Time Frame: From baseline to 31 months
Population: FAS population with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 22 | 29 | 9
Scores on scale | 0.77 (3.98) | 0.87 (2.92) | 1.37 (3.49)
Statistical Analysis 1: Comparison: Randomized Cohort: Gilteritinib + AZA vs Randomized Cohort: AZA; Test type: Superiority; p = 0.560, ANCOVA; Using analysis of covariance including treatment, age group per IRT and baseline score as covariate; Least square mean difference = 0.5, 95% CI 2-sided [-1.1 to 2.0] — Least square mean difference and P-value were calculated using AZA as reference

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE was defined as an adverse event observed after starting administration of the study drug until 30 days from the last study treatment
Time Frame: From first dose up to end of study duration (101 months)
Population: The Safety Analysis Set (SAF) consisted of all participants who received at least one dose of study drug (ASP2215 or azacitidine).
Measure: Number; unit: participants
Groups:
- Safety Cohort: Gilteritinib + AZA: Participants received 80 mg (2 tablets of 40 mg) of gilteritinib orally once daily for continuous 28-day cycles and 75 mg/m^2 of AZA daily via subcutaneous injection or intravenous infusion for 7 days of each 28-day treatment cycle. Depending on the safety cohort data ,the decision to initiate the randomized trial at the targeted dose was made.
Arm/Group | Safety Cohort: Gilteritinib + AZA | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 15 | 88 | 54 | 22
participants | 15 | 88 | 52 | 22

14. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Scores
Description: ECOG performance scores at each assessment time were be provided by treatment group. Negative change scores indicated an improvement and positive scores indicate a decline in performance. The grades were defined as follows:
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Time Frame: From baseline to end of treatment (up to 57 months)
Population: SAF population with available data was analyzed.
Measure: Number; unit: participants
Arm/Group | Safety Cohort: Gilteritinib + AZA | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
Number analyzed (Participants) | 15 | 88 | 54 | 22
participants
  Baseline: Grade 0 | 1 | 15 | 9 | 3
  Baseline: Grade 1 | 4 | 34 | 26 | 6
  Baseline: Grade 2 | 4 | 28 | 14 | 9
  Baseline: Grade 3 | 6 | 10 | 5 | 3
  Baseline: Grade 4 | 0 | 1 | 0 | 1
  Baseline: Grade 5 | 0 | 0 | 0 | 0
  End of Treatment (EOT): Grade 0: number analyzed (Participants) | 6 | 41 | 36 | 11
  End of Treatment (EOT): Grade 0 | 1 | 4 | 8 | 2
  EOT: Grade 1: number analyzed (Participants) | 6 | 41 | 36 | 11
  EOT: Grade 1 | 1 | 12 | 15 | 4
  EOT: Grade 2: number analyzed (Participants) | 6 | 41 | 36 | 11
  EOT: Grade 2 | 2 | 12 | 11 | 3
  EOT: Grade 3: number analyzed (Participants) | 6 | 41 | 36 | 11
  EOT: Grade 3 | 1 | 7 | 1 | 1
  EOT: Grade 4: number analyzed (Participants) | 6 | 41 | 36 | 11
  EOT: Grade 4 | 1 | 6 | 1 | 1
  EOT: Grade 5: number analyzed (Participants) | 6 | 41 | 36 | 11
  EOT: Grade 5 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): From randomization up to end of study duration (101 months) AEs: From first dose up to end of study duration (101 months)
Description: ACM: All randomized participants.
  AEs: SAF consisted of all participants who received at least one dose of study drug (ASP2215 or azacitidine).
Arm/Group | Safety Cohort: Gilteritinib + Azacitidine (AZA) | Randomized Cohort: Gilteritinib + AZA | Randomized Cohort: AZA | Randomized Cohort: Gilteritinib
All-Cause Mortality (participants affected / at risk) | 14/15 | 70/89 | 49/57 | 22/22
Serious Adverse Events (participants affected / at risk) | 14/15 | 81/88 | 34/54 | 20/22
Other Adverse Events (participants affected / at risk) | 15/15 | 87/88 | 46/54 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Cohort: Gilteritinib + Azacitidine (AZA) (N=15) | Randomized Cohort: Gilteritinib + AZA (N=88) | Randomized Cohort: AZA (N=54) | Randomized Cohort: Gilteritinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 4 (5) | 0 (0) | 2 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (16) | 28 (49) | 10 (12) | 4 (10)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 1 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 7 (9) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinitis pigmentosa (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acquired macroglossia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (7) | 12 (21) | 1 (1) | 5 (6)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (7) | 19 (28) | 8 (9) | 5 (9)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 9 (13) | 5 (9) | 4 (6)
Septic embolus (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 6 (11) | 1 (1) | 5 (6)
Soft tissue infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 6 (7) | 0 (0) | 3 (4)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 4 (5) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Cohort: Gilteritinib + Azacitidine (AZA) (N=15) | Randomized Cohort: Gilteritinib + AZA (N=88) | Randomized Cohort: AZA (N=54) | Randomized Cohort: Gilteritinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 8 (13) | 28 (59) | 18 (30) | 6 (10)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (8) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (23) | 28 (104) | 16 (35) | 3 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (12) | 29 (63) | 11 (14) | 4 (11)
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (7) | 3 (3) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 35 (52) | 13 (16) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 30 (53) | 10 (12) | 9 (12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (2) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 6 (6) | 3 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 8 (8) | 2 (2) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (10) | 27 (55) | 13 (13) | 3 (3)
Oral pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 6 (7) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (8) | 23 (38) | 10 (10) | 7 (8)
Asthenia (General disorders) | 2 (3) | 20 (37) | 9 (10) | 2 (4)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (13) | 8 (10) | 5 (7) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Injection site erythema (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 5 (6) | 3 (4) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Oedema (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (5) | 26 (43) | 8 (9) | 7 (8)
Pain (General disorders) | 1 (2) | 4 (5) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 37 (79) | 17 (18) | 5 (12)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 4 (6) | 0 (0) | 2 (2)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 8 (9) | 1 (1) | 1 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 5 (6) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 9 (9) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 7 (7) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 10 (15) | 5 (5) | 3 (3)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 1 (2) | 6 (7) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 6 (8) | 5 (8) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (8) | 3 (4) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8) | 15 (47) | 5 (6) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 19 (56) | 3 (3) | 4 (9)
Blood alkaline phosphatase increased (Investigations) | 2 (4) | 9 (14) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 6 (7) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 8 (19) | 0 (0) | 2 (6)
Blood creatinine increased (Investigations) | 4 (4) | 15 (27) | 3 (4) | 6 (10)
Blood glucose increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (2) | 2 (5) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 8 (18) | 0 (0) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 5 (10) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 14 (91) | 4 (5) | 2 (8)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (7) | 15 (45) | 9 (22) | 6 (44)
Transaminases increased (Investigations) | 0 (0) | 6 (12) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 9 (9) | 4 (4) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 8 (48) | 3 (5) | 3 (12)
Decreased appetite (Metabolism and nutrition disorders) | 4 (7) | 16 (25) | 10 (12) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (9) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (9) | 1 (1) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (8) | 1 (1) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 7 (14) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 14 (25) | 1 (1) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (5) | 11 (16) | 2 (4) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 22 (48) | 10 (15) | 4 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 10 (32) | 3 (3) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 15 (28) | 4 (4) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 12 (37) | 3 (3) | 3 (4)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (17) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (3) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 5 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (12) | 3 (4) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 7 (12) | 4 (4) | 4 (7)
Headache (Nervous system disorders) | 2 (3) | 7 (12) | 3 (4) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 3 (3) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 9 (13) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 14 (16) | 3 (4) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 6 (7) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 5 (7) | 3 (4) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 3 (5) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 5 (6) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (11) | 3 (4) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 11 (17) | 4 (5) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 12 (17) | 5 (6) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (11) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8) | 2 (2) | 3 (3)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (16) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (13) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 5 (5) | 2 (5)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (2) | 9 (9) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (3) | 9 (12) | 2 (4) | 2 (2)
Hypotension (Vascular disorders) | 3 (4) | 12 (14) | 3 (6) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Protocol versions 6.0 and earlier included a 1:1:1 randomization ratio to receive Gilteritinib + AZA, AZA-only and Gilteritinib-only. Randomization to arm Gilteritinib-only was removed in protocol version 7.0. Participants previously randomized to Gilteritinib-only arm continued following treatment and assessments as outlined in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT02752035/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT02752035/SAP_001.pdf